CLINICAL TRIAL: NCT05436041
Title: Pilot Trial of Nutri, a Clinical Decision Support Software to Improve Diet Goal-Setting in Primary Care
Brief Title: Nutri Diet Goal Setting Software Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Lone Star Circle of Care (Unknown)
Responsible Party: Principal Investigator, Marissa Burgermaster, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 201903265; 1R21HS027660 (AHRQ)
Record Dates: First submitted 2022-06-10; First posted 2022-06-28 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes; Pre-diabetes; Metabolic Syndrome
Keywords: Clinical Decision Support; Dietary Management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutri (Experimental): PCPs will receive an alert to use Nutri personalized diet goal setting software with enrolled patients
  Interventions: Behavioral: Collaborative Diet Goal Setting Clinical Decision Support
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Collaborative Diet Goal Setting Clinical Decision Support — Receives Nutri
  Other Names: Nutri
  Arms: Nutri

SUMMARY:
The investigators will conduct a pilot cluster randomized trial of Nutri, a clinical decision support software to support collaborative diet goal setting in primary care. Nutri is designed within the Chronic Care Model framework, specifically with the intention of leveraging clinical information systems to connect clinical care with patients' lives in the community setting. Nutri is based on the Theory of Planned Behavior and uses collaborative goal setting between the patient and provider to identify a behavioral intention (i.e., diet goal) and improve goal self-efficacy by improving attitudes/outcome expectations, subjective norms/social support, and perceived behavioral control.

In this pilot trial, the intervention group (N=10 primary care providers [PCPs], N=40 patients) receives collaborative diet goal setting via Nutri, and the control group receives usual care(N=10 PCP, N=40 patients). Before and after the appointment, patients will report food they consumed over the last 24 hours via the dietary recall tool, ASA24 and respond to surveys about behavioral intention and self-efficacy. Intervention PCPs will be alerted when the Nutri workflow is available for a patient and asked to complete it during their visit with that patient.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Diagnosed with pre-diabetes or type 2 diabetes, or at risk for type 2 diabetes
3. Have a scheduled medical appointment with a study enrolled PCP within the study enrollment period
4. Fluent in either English or Spanish
5. Access to a computer, tablet, or smartphone and reliable internet
6. Stated willingness to comply with all study procedures and availability for the duration of the study
7. HIPAA authorization for Health Information Exchange

Exclusion Criteria:

1. Currently pregnant
2. Diagnosed with an eating disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Variance and Within-Provider Covariance of Patient Self-Reported Dietary Behavioral Intention | 1-day post medical encounter
  Patient self-report of a diet goal set during medical appointment, coded y/n
Variance and Within-Provider Covariance of Patient Self-Reported Dietary Behavior Change Self-Efficacy (Confidence in ability to change dietary behavior) | 1-day post medical encounter
  Patient self-report of self-efficacy (ie, confidence) in changing their diet after appointment, 7-point Likert scale, a higher score means a better outcome
Variance and Within-Provider Covariance of Patient Change in Diet Quality (measured via Healthy Eating Index) | Patient pre-assessment and 7-day post medical encounter
  Change in diet quality measured via the Healthy Eating Index (HEI) score calculated from 24-hour recall, 0-100 score range, higher score means better outcome.

SECONDARY OUTCOMES:
Nutri (Intervention) Usability | PCP post-assessment (after 4 medical encounters), expected to be at 8 weeks after enrollment
  System Usability Scale, 0-100 score range, higher score means better outcome
Number and timeline of PCPs and patients recruited into the study | through study completion, expected to be at 8 weeks after enrollment
  Recruitment of patients and providers into the study, including timeline and total number. The outcome will be used to inform pragmatic trial feasibility.
Number and timeline of PCPs and patients who drop out of the study | through study completion,expected to be at 8 weeks after enrollment
  Loss to follow up of patients and providers into the study, including timeline and total number. The outcome will be used to inform pragmatic trial feasibility.
Completion of patient ASA24 survey | patient pre-assessment & 7 days post-appointment
  Patient completion of the ASA24 survey pre and post-test. The outcome will be used to inform pragmatic trial feasibility.
Impact of Nutri on Patient Self-Reported Dietary Behavioral Intention | 1 day post-medical encounter
  Difference between intervention and control in the frequency of patient self-reported diet goal.
Impact of Nutri on Patient Self-Reported Dietary Behavior Change Self-Efficacy (Confidence in ability to change dietary behavior), measured via questionnaire | 1 day post-medical encounter
  The difference between intervention and control in the amount of patient self-reported self-efficacy (confidence) in changing their diet after the appointment, 7-point Likert scale, a higher score means a better outcome.
Impact of Nutri on Patient Diet Quality (measured via Healthy Eating Index) | Patient pre-assessment and 7 days post-medical encounter
  Difference between intervention and control in change in Healthy Eating Index (HEI) score calculated from 24-hour recall, 0-100 score range, a higher score means a better outcome.

OTHER OUTCOMES:
Impact of Nutri on PCP Diet Counseling Self-Efficacy | PCP pre-assessment and PCP post-assessment (after 4 medical encounters), expected to be at 8 weeks after enrollment
  PCP self-report of confidence (self-efficacy) in diet counseling; 4-point likert scale; higher score means better outcome
Impact of Nutri on PCP Attitude Toward Diet Counseling. | PCP pre-assessment and PCP post-assessment (after 4 medical encounters), expected to be at 8 weeks after enrollment
  PCP self-report of attitude towards diet counseling; 4-point Likert scale; higher score means better outcome
Impact of Nutri on PCP Diet Counseling Competency | PCP pre-assessment and PCP post-assessment (after 4 medical encounters), expected to be at 8 weeks after enrollment
  PCP self-report of diet counseling competency; 4-point likert scale; higher score means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Marissa Burgermaster, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- Lone Star Circle of Care, Austin, Texas, United States